CLINICAL TRIAL: NCT04650269
Title: Implementation of Onsite, Rapid Antiretroviral Therapy (ART) Initiation Among People Who Inject Drugs Living With HIV at Syringe Services Program
Brief Title: Implementation of Onsite, Rapid ART Initiation Among People Who Inject Drugs Living With HIV at Syringe Services Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Hansel Tookes, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200793
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Harm Reduction; HIV Infections; Drug Use
MeSH Terms: conditions — Harm Reduction; HIV Infections | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rapid ART group (Experimental): Patients will receive HIV care including Biktarvy for 6 months at the syringe services program followed by 6 months of standard of care at a traditional clinic.
  Interventions: Drug: Biktarvy 50Mg-200Mg-25Mg Tablet; Other: HIV care

INTERVENTIONS:
Drug: Biktarvy 50Mg-200Mg-25Mg Tablet — Daily Biktarvy (50/200/25mg) combination ART by mouth for 6 months
Other: HIV care — HIV primary care (including Biktarvy delivery) will be conducted outside of a clinical setting by a community-based harm reduction program for 6 months.

SUMMARY:
The purpose of this study is to see if providing HIV medicine right away at the IDEA Syringe Services Program will help the participant start and remain in HIV care, including having no detectable HIV in the participant's blood.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age>18 years);
2. positive rapid HIV test;
3. ability to provide informed consent;
4. HIV RNA > 200 copies/ml;
5. creatinine clearance > 30 mg/dl as measured by serum creatinine;
6. no allergy to bictegravir/emtricitabine/tenofovir alafenamide (BFTAF) as indicated by patient history and self-reported allergies.

Exclusion Criteria:

1) Any other comorbidities at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation
Enrollment: 27 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hansel Tookes, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rapid ART Group
Started | 27
Completed | 18
Not Completed | 9
Not completed — Death | 3
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Rapid ART Group
Number analyzed (Participants) | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [34 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV Viral Load Suppression
Description: HIV viral load suppression is defined as <200 copies/ml in participants' blood
Time Frame: 6 months
Population: Data was not collected for those participants that were lost to follow-up or death due to COVID pandemic
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid ART Group
Number analyzed (Participants) | 16
Participants | 11

2. Secondary Outcome: Percentage of Participants With HIV Viral Load Suppression
Description: HIV viral load suppression is defined as <200 copies/ml in participants' blood
Time Frame: 1 month
Population: Data was not collected for those participants that were lost to follow-up or death due to the COVID pandemic
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid ART Group
Number analyzed (Participants) | 16
Participants | 11

3. Secondary Outcome: Percentage of Participants With HIV Viral Load Suppression
Description: HIV viral load suppression is defined as <200 copies/ml in participants' blood
Time Frame: 12 months
Population: Data was not collected for those participants that were lost to follow-up or death due to the COVID pandemic
Measure: Count of Participants; unit: Participants
Arm/Group | Rapid ART Group
Number analyzed (Participants) | 19
Participants | 15

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Rapid ART Group
All-Cause Mortality (participants affected / at risk) | 3/27
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapid ART Group (N=27)
death (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/69/NCT04650269/Prot_SAP_000.pdf